CLINICAL TRIAL: NCT03930407
Title: Serum Antimullerian Hormone Levels in Patients Who Underwent Hayman Suture for Uterine Atony During Cesarean Section
Brief Title: Serum Antimullerian Hormone Levels in Patients Who Underwent Hayman Suture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aysu Akca, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: AYSUAKCA1
Record Dates: First submitted 2019-04-23; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Uterine Atony With Hemorrhage; Ovarian Dysfunction
Keywords: Cesarean section; Uterine atony; Hayman uterine compression suture; Follicle-stimulating hormone; Luteinizing hormone; Antral follicle count
MeSH Terms: conditions — Uterine Inertia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hayman group: Who had undergone cesarean section within the last 6 months and received a The Hayman uterine compression suture for uterine atony.
  Interventions: Procedure: The Hayman uterine compression suture.
- Control: Who had undergone cesarean section within the last 6 months and did not experience neither any complication nor any additional intervention

INTERVENTIONS:
Procedure: The Hayman uterine compression suture. — Hayman suture is a common technique for uterine compression to stop bleeding due to uterine atony. Hayman described placement of two to four vertical compression sutures from the anterior to posterior uterine wall without hysterectomy. It is usually employed to overcome uterine atony during cesarean section.
  Groups: Hayman group

SUMMARY:
From patient charts we will review patients who had undergone cesarean section within the last 6 months and identify those who received a The Hayman uterine compression suture for uterine atony. We will also select patients who delivered a baby without recieving a Hayman suture to create a control group. Patietns will be grouped as Hayman Group if they recevied a Hayman suture during C/S and control group if thay had not recevied a Hayman suture. We will then check patient charts for post-cesarean outpatient clinic visit and select those who received ovarian reserve evaluation via hormones and antral follicle count during the visits. Finally, we are planning to investigate any correlation between Hayman suture and ovarian dysfunction.

DETAILED DESCRIPTION:
Hayman suture is a common technique for uterine compression to stop bleeding due to uterine atony. Hayman described placement of two to four vertical compression sutures from the anterior to posterior uterine wall without hysterectomy. It is usually employed to overcome uterine atoy dıring cesarean section. However, since the technique is relatively new, data on its safety and efficacy arelimited to a few case reports. several complications including cavity obliteration, blood entrapment and infections have been described. However, data regarding the ovarioan function is lacking.

ELIGIBILITY:
Inclusion Criteria:

* age 18- 40 years
* no systemic or endocrine diseases
* patients who had uterine artery ligation due to atony
* healthy postpartum patients as controls

Exclusion Criteria:

* patients with Polyctsitic over syndrome
* Pregnancy with IVF or oocyte donation
* Obese patients
* patients with previous/present endometriosis

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Patients who had undergone uterine artery ligation during cesarean section. Control group is age-matched postpartum patients.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-06-10 (Estimated); Study Completion 2019-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in anti-mullerian hormone level from baseline (precesarean) to post-cesarean | Before cesarean section and at any follow-up visit within 6 months of cesarean section
  ng/dl
Change in follicle stimulating hormone level from baseline (precesarean) to post-cesarean | Before cesarean section and at any follow-up visit within 6 months of cesarean section
  IU/L
Change in luteinizing hormone level from baseline (precesarean) to post-cesarean | Before cesarean section and at any follow-up visit within 6 months of cesarean section
  mU/mL

SECONDARY OUTCOMES:
Antral follicle count in the two study groups | At any follow-up visit within 6 months of cesarean section
  number

CONTACTS AND LOCATIONS:
Overall Officials: Asyu Akca, Principal Investigator — Kanuni Sultan Suleyman Hospital
Locations (1):
- Department of Obstetrics and Gynecology, University of Health Sciences, Faculty of Medicine, Kanuni Sultan Suleyman Hospital,, Istanbul, Please Enter the State Or Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided